CLINICAL TRIAL: NCT03305679
Title: Evaluation of the Clinical Efficacy of the Immediate Implant Loading in the Aesthetic Zone
Brief Title: Clinical Efficacy of the Immediate Implant Loading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Collaborators: St Joseph University, Beirut, Lebanon (Other); Syrian Atomic Energy Agency, Damascus, Syria (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UDDS-FixPro-01-2017
Record Dates: First submitted 2017-10-02; First posted 2017-10-10 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Implant Site Reaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct provisional technique (Experimental): Patients here will be subjected to the direct provisional technique
  Interventions: Procedure: Direct provisional technique
- Indirect Provisional technique (Active Comparator): Patients here will be subjected to the indirect provisional technique
  Interventions: Procedure: Indirect Provisional technique

INTERVENTIONS:
Procedure: Direct provisional technique — The method of implantation will be accomplished directly.
  Arms: Direct provisional technique
Procedure: Indirect Provisional technique — The method of implantation will be accomplished indirectly.
  Arms: Indirect Provisional technique

SUMMARY:
Aim: The aim of this study to Assess the healing process of the immediate implant loading with two different provisional techniques (direct and indirect).

Materials and methods:

20 implant in the aesthetic zone either in the incisor or in the canine area and excluding the lateral location and then immediate loading is achieved for the 20 implants (10 for direct and 10 for indirect method) Clinical Aspect :color change , healing and bone resorption Esthetic assessment and patient acceptance will be assessed using specific tools.

Lab aspect: surface roughness and Marginal fit will be measured to have clue vision.

DETAILED DESCRIPTION:
Aim: The aim of this study to Assess the healing process of the immediate implant loading with two different provisional techniques (direct and indirect).

Materials and methods:

20 implant (Implant Direct ) in the aesthetic zone either in the incisor or in the canine area and excluding the lateral location and then immediate loading is achieved for the 20 implants (10 for direct and 10 for indirect method) Clinical Aspect :color change , healing and bone resorption Aesthetic assessment and patient acceptance will be assessed using specific tools Lab aspect: surface roughness and Marginal fit will be measured to have clue vision.

The participants were non-dental students from University colleges in and around Damascus. They were recruited by reviewing the case documents 20 patient with hapless incisal and canine for extraction and immediate implantation and immediate loading with either the two different provisional methods participants had to demonstrate a hopeless central incisor or canine with no perio-active infection. With two types of provisional technique we will have a two groups were calculated a priori in such a way that index can be identified with with alpha = .05 in a two-tailed test, a sample size of 2 X10 implants would result in a power of 94% (g power 3.1.3) based on a pilot study.

Cone-beam computed tomography (CBCT) images for each patient to measure the bone level change and aesthetic assessment by three general dentists will be achieved. Replica technique required the application of impression material build up of addition-silicone. Addition-silicone of very low viscosity (ExpressTM2 Ultra-Light Body Quick) was applied to all restorations interior, after which the crowns were set onto basic samples. Impression material was polymerized within the time which is recommended by the manufacturer, while the pressure force of 50 N was applied toward occlusal direction After the removal of all restorations from the basic samples, the layer of impression material remained on the restoration's inner surface due to its higher roughness compared to the abutment surface. With Rt 200 device the roughness will bw measured and then Scanning Electronic Microscope (SEM) images will give a close understanding of the surface. Easy shade will measure the color change.

ELIGIBILITY:
Inclusion Criteria:

1. esthetic request.
2. either incisor or canine indicated for extraction.
3. symmetrical gingival level.
4. no active periodontal disease.
5. age between 20-40 years old

Exclusion Criteria:

1. Lateral hopeless tooth .
2. Active periodontal lesion .
3. loss of periodontal tissue .
4. missed incisor or missed canine in the area of implantation.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-07-19 (Actual)

PRIMARY OUTCOMES:
Change in alveolar bone level | T1: at one day after implantation, T2: at one month following implantation, T2: at two months following implantation, T3: at three months following implantation
  This will be measured using cone-beam computed tomography images
Change in the Gingival Index | T1: at one day after implantation, T2: at one month following implantation, T2: at two months following implantation, T3: at three months following implantation
  This will be measured using the the gingival index
Change in Esthetic Appearance | T1: at one day before implantation, T2: at three months following implantation
  This will be measured by using the White Esthetic Scale (WES)
Change in the Plaque Index | T1: at one day after implantation, T2: at one month following implantation, T2: at two months following implantation, T3: at three months following implantation
  This will be measured using the the plaque index
Change in the Pink Esthetic Scale | T1: at one day after implantation, T2: at one month following implantation, T2: at two months following implantation, T3: at three months following implantation
  This will be measured using the Pink Esthetic Scale

SECONDARY OUTCOMES:
Change in Restoration Color | T1: at one day after implantation, T2: at one month following implantation, T2: at two months following implantation, T3: at three months following implantation
  This will be measured using a standardized color guide

CONTACTS AND LOCATIONS:
Overall Officials: Anas Abdo, DDS MSc, Principal Investigator — PhD student in Fixed Prosthodontics, Department of Fixed Prosthodontics, University of Damascus Dental School; Osama Yousuf Solieman, DDS MSc PhD, Study Director — Laboratoire Bioinge Ânierie et Nanosciences EA4203, Montpellier University, Montpellier, France; Christian Makary, DDS MSc PhD, Study Director — Professor of Oral Implantology, Sante Jousef University, School of Dental Medicine, Beirut, Lebanon; Mirza Allaf, DDS MSc PhD, Study Chair — Professor of Fixed Prosthodontics, University of Damascus Dental School, Damascus, Syria
Locations (3):
- Department of Oral Implantology -Sante Jousef University - School of Dental Medicine, Beirut, Lebanon
- Syria (2):
  - Department of Fixed Prosthodontics, University of Damsacus, Damascus
  - Nano Physical lab and biomaterial Lab - College of Applied Sciences, Damascus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friberg B. Bone augmentation for single tooth implants: A review of the literature. Eur J Oral Implantol. 2016;9 Suppl 1:S123-34. PMID 27314117
- [Background] Sanchez-Siles M, Munoz-Camara D, Salazar-Sanchez N, Camacho-Alonso F, Calvo-Guirado JL. Crestal bone loss around submerged and non-submerged implants during the osseointegration phase with different healing abutment designs: a randomized prospective clinical study. Clin Oral Implants Res. 2018 Jul;29(7):808-812. doi: 10.1111/clr.12981. Epub 2016 Sep 5. PMID 27596682
- [Background] Stoupel J, Lee CT, Glick J, Sanz-Miralles E, Chiuzan C, Papapanou PN. Immediate implant placement and provisionalization in the aesthetic zone using a flapless or a flap-involving approach: a randomized controlled trial. J Clin Periodontol. 2016 Dec;43(12):1171-1179. doi: 10.1111/jcpe.12610. Epub 2016 Oct 17. PMID 27501953
- [Background] Sethi A, Kaus T. Immediate Replacement of Single Teeth With Immediately Loaded Implants: Retrospective Analysis of a Clinical Case Series. Implant Dent. 2017 Feb;26(1):30-36. doi: 10.1097/ID.0000000000000512. PMID 27902498
- [Background] Zhang S, Wang S, Song Y. Immediate loading for implant restoration compared with early or conventional loading: A meta-analysis. J Craniomaxillofac Surg. 2017 Jun;45(6):793-803. doi: 10.1016/j.jcms.2016.05.002. Epub 2016 May 14. PMID 28351528
- [Background] Abdel-Azim T, Rogers K, Elathamna E, Zandinejad A, Metz M, Morton D. Comparison of the marginal fit of lithium disilicate crowns fabricated with CAD/CAM technology by using conventional impressions and two intraoral digital scanners. J Prosthet Dent. 2015 Oct;114(4):554-9. doi: 10.1016/j.prosdent.2015.04.001. Epub 2015 Jun 20. PMID 26100929
- [Background] Varol S, Kulak-Ozkan Y. In Vitro Comparison of Marginal and Internal Fit of Press-on-Metal Ceramic (PoM) Restorations with Zirconium-Supported and Conventional Metal Ceramic Fixed Partial Dentures Before and After Veneering. J Prosthodont. 2015 Jul;24(5):387-93. doi: 10.1111/jopr.12229. Epub 2014 Oct 1. PMID 25274041
- [Background] Renne W, Wolf B, Kessler R, McPherson K, Mennito AS. Evaluation of the Marginal Fit of CAD/CAM Crowns Fabricated Using Two Different Chairside CAD/CAM Systems on Preparations of Varying Quality. J Esthet Restor Dent. 2015 Jul-Aug;27(4):194-202. doi: 10.1111/jerd.12148. Epub 2015 Jul 14. PMID 26177118
- [Background] Louropoulou A, Slot DE, Van der Weijden F. Influence of mechanical instruments on the biocompatibility of titanium dental implants surfaces: a systematic review. Clin Oral Implants Res. 2015 Jul;26(7):841-50. doi: 10.1111/clr.12365. Epub 2014 Mar 19. PMID 24641774